CLINICAL TRIAL: NCT00002403
Title: A Phase I/II Multiple Dose Study to Evaluate the Safety, Pharmacokinetic Profile and Virologic/Immunologic Activity of Zintevir (AR177) in HIV-1 Patients
Brief Title: Safety and Effectiveness of Zintevir (AR177) Given to HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aronex Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 290A; UNAP 3; AR177-003
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-12

CONDITIONS: HIV Infections
Keywords: HIV-1; Dose-Response Relationship, Drug; HIV Integrase Inhibitors; HIV Integrase
MeSH Terms: conditions — HIV Infections | interventions — T 30177

INTERVENTIONS:
Drug: Zintevir

SUMMARY:
The purpose of this study is to see if it is safe and effective to give zintevir (AR177) to asymptomatic (no symptoms) HIV-infected patients.

Zintevir belongs to a new class of anti-HIV drugs, the integrase inhibitors. HIV uses the protein integrase to infect a cell. Integrase inhibitors block integrase and may stop replication of HIV.

DETAILED DESCRIPTION:
Zintevir belongs to a new class of anti-HIV drugs, the integrase inhibitors. The HIV-1 virus uses the protein integrase to incorporate its genetic material into the infected host cell. Integrase inhibitors block integrase and may stop replication of the HIV-1 virus.

In this open-label, Phase I/II study, 3 groups of HIV-positive patients (12 patients total) receive escalating doses of intravenous zintevir for 14 consecutive days.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive, but do not have any symptoms of HIV infection.
* Have a CD4 count greater than 200 cells/mm3.
* Have a viral load (level of HIV in the body) greater than 4,000 copies/ml.
* Are at least 18 years old.

Exclusion Criteria

You will not be eligible for this study if you:

* Tend to have abnormal bleeding or other blood problems.
* Have an active AIDS-defining illness.
* Have a history of serious disease or illness.
* Abuse alcohol or drugs.
* Have received certain medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12

CONTACTS AND LOCATIONS:
Locations (1):
- Cornell AIDS Clinical Trials Unit, New York, New York, United States